

**Unique Protocol ID:** Nu-V3 Phase I **NCT Number:** (not yet assigned)

Brief Title: Nu-V3 Non-Invasive Nerve Stimulation Device Trial for Pain,

Anxiety, Depression, Sleeplessness

**Official Title:** A Phase I Prospective, Single-Arm, Open-Label, Multi-Center Study Using the Nu-V3 Cranial Nerve Stimulation Treatment Device in Patients With Pain, Anxiety, Depression, and/or Sleeplessness

INVESTIGATIONAL DEVICE: Nu-V3 SPONSOR: Nu-Life Solutions

# Phase I & II Statistical Analysis Plan\*

\*\*All initial graphs and table data are simulated and will be updated at time of study submission

VERSION DATE: 03/APR/2018



## **Summary of Clinical Information**

The primary pivotal study provided to support the De Novo request is the "Nu-V3 Protocol No. 1"- phases I & II. Details of the study design and selected clinical results are provided below.

**Purpose:** The objective of this research study was to collect data which demonstrates the ability of the Nu-V3 device to offer relief from one or more of the following symptoms: pain, depression, anxiety, and/or sleeplessness. The objective is to demonstrate the effectiveness of Nu-V3 for any or all of the four symptoms listed.

| Design: The Nu-V3 ( | Clinical Study was a p | prospective, single-arm, open-label, multi-center, |
|---|---|---|
| global study using the | e Nu-V3 cranial nerve | stimulation treatment device in patients with |
| uncontrolled pain, an | xiety, depression, and | d/or sleeplessness. For the Phase I study, a total of |
| patients at | centers in the | e United States were registered for study participation |
| A total of | patients at | centers in the United States, Japan, India, |
| Germany, United Kin | gdom, Austria, Switze | erland, , were registered to the Phase II |
| study. | | • |

**Phase I study** consisted of 50-100 individuals who signed the informed consent form, met the inclusion and exclusion criteria, and were enrolled in the study at multiple sites. Enrolled participants are treated with the Nu-V3 device for 8 weeks, then observed for an additional 2 weeks. Interim analysis of reported data were conducted at 4, 8, and 12 weeks during this time. Post study, participants were given the chance to continue with an optional maintenance treatment with the Nu-V3 device per a 2-week on, 2-week off schedule, for an additional 12 weeks, with an 8-week observation.

**Phase II of the study** consisted of 100-200 individuals who signed the informed consent form, met the inclusion and exclusion criteria, and were enrolled in the study at multiple sites. Enrolled participants are treated with the Nu-V3 device for 8 weeks, then observed for an additional 2 weeks. Interim analysis of reported data were conducted at 4, 8, and 12 weeks during this time. Post study, participants were given the chance to continue with an optional maintenance treatment with the Nu-V3 device per a 2-week on, 2-week off schedule, for an additional 12 weeks, with an 8-week observation.

Subjects enrolled onto the Nu-V3 Clinical Trial underwent the following regimen:

- At the baseline visit, patients will be asked to complete study questionnaires regarding all of the following symptoms: pain, depression, anxiety, and/or sleeplessness, as well as their activity level, active medications, and demographics information.
- At each subsequent visit, patients will be asked to complete study questionnaires regarding all the following symptoms: pain, depression, anxiety, and/or sleeplessness, as well as their activity level.
- The sessions will begin with the Nu-V3 device being placed on the ear and three small pads (non-invasive) being placed on the ear. Each Nu-V3 device lasts for up to 14 days with a change in the pads approximately 7 days into the treatment.
- Each session takes approximately 15-20 minutes. The placement of the device takes approximately 5 minutes and the remaining time is spent verifying assessment form completion and checking for any immediate effects from the device.
- The Nu-V3 device is mobile and is worn externally on the ear 24 hours a day during treatment, fitting comfortably behind the ear. An electrical signal is sent to the external



ear through coated wire leads attached to the device and adhesive pads which attach to three sites on the ear.

- Participants should be able to perform their typical day-to-day activities while wearing
  the device. They may shower while wearing the Nu-V3 device, provided that they do not
  get the device wet and use the small disposable ear covers that are provided for them.
- Patients should not change their existing forms of treatment or medications without discussion with the investigator.
- Nu-Life reserves the right to capture video, photographs and written testimonials from
  patients with written permission. In the event subjects elect to participate in any or all of
  these activities, they will be asked to sign a waiver giving exclusive rights to the video,
  photographs and written testimonials captured to Nu-Life. Their participation in this study
  is not dependent upon their willingness to participate in video, photographs or written
  testimonials.

| | | | | Stu | idy T | reatm | ent | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Evaluation* | | Week<br>2 | Week<br>3 | Week<br>4 | Week<br>5 | Week<br>6 | Week<br>7 | Week<br>8 | Week<br>9-11 | Week |
| Informed Consent | x | | | | | | | | | |
| Inclusion and Exclusion <sup>1</sup> | X | | | | | 3 | | | | |
| Patient Registration <sup>1</sup> | х | | | | | | | | | |
| Medications Form <sup>1</sup> | х | S | | х | FG - X2 | | | х | | х |
| Patient Onboarding and Orientation <sup>2</sup> | х | 3 0) | | | | | | | | |
| In office assessment | х | х | x | х | х | x | x | х | 3 | × |
| New Device Placed | × | 8 03 | x | | х | | х | | | |
| Pad Replaced | | х | | х | | x | | х | | |
| Treatment Forms <sup>1</sup> | х | х | х | х | х | х | х | х | | |
| No Device | | R X | 2 | | 70 XX | 2 | | | х | х |
| ePRO Questionnaires <sup>3</sup> | х | х | х | х | х | х | х | х | х | х |
| Patients' Global Impression of Change ePRO form (PGIC) <sup>3</sup> | | х | x | х | х | х | x | х | - 3 | х |
| Providers' Global Impression of Change ePRO form (PGIC) | | х | x | X | х | x | х | х | | х |
| Family Global Impression of Change ePRO form (PGIC) | | x | х | x | х | x | x | x | | x |
| Optional Patient Media Testimony | х | | | х | 1 | | | x | 1 | х |

- 12. Inclusion/Exclusion, Registration, Medications, Treatment forms to be completed by site coordinator via online module.
- 2. Patient Onboarding and Orientation includes introductory demographics form, Nu-V3 patient training video
- 3. ePRO questionnaires completed on patient's mobile device: DQ-9 (baseline), PTB-7, PEG, GAD-7, PHQ-9, PROMIS 4a, PGIC
- 4. If patient consents to media testimony, site will collect via study collection process every 4 weeks.

**Study Endpoints and Data Analysis:** The study endpoints data were collected from each participant's study questionnaires. The data were collected electronically via the patient's own device, and were uploaded to an electronic data capture system. The data were used to demonstrate that the Nu-V3 device provides participants with relief of the symptoms of pain, depression, anxiety and/or sleeplessness. The data analysis includes comparative data for each participant's questionnaire prior to beginning treatment with the Nu-V3 device, the participant's weekly questionnaires during treatment and the questionnaire completed at the end of the treatment with the Nu-V3 device.



### **Primary Endpoints:** Primary endpoints consisted of the following:

- 1. <u>Safety</u>: The primary safety endpoint was the occurrence of reported unanticipated problems involving risk to subjects or others ("UPIRTSOs"). These UPIRTSOs are defined as those problems which alter the risks to subjects or others. This includes any study suspensions or holds. The primary safety endpoint analyses were based on a risk-benefit conclusion.
- 2. Effectiveness: The primary effectiveness endpoints were overall reduction in median reported symptoms of pain, anxiety, depression, and/or sleeplessness via numeric rating scales at 8 weeks. This primary effectiveness is measured by median reported symptom reductions in pain, anxiety, depression, and/or sleeplessness via the following validated tools: Pain intensity and interference- PEG Scale, Anxiety- Generalized Anxiety Disorder 7-item (GAD-7) scale, Depression- Patient Health Questionnaire (PHQ-9), Sleeplessness-PROMIS short form 4a, and overall improvement of quality of life (QOL) Patient's Global Impression of Change (PGIC).

The patient's perceived treatment benefit and device comfort information, will be captured via the non-validated tool, Perceived Treatment Benefit Form (PTB-7). This effectiveness tool will measure median levels of reported perceived treatment benefit and device comfort.

The hypothesis-driven criterion of effectiveness was to show that there was a statistically significant reduction in the median reported pain, anxiety, depression, and/or sleeplessness levels of patients using the Nu-V3 device. The second criterion was intended to show that there was a statistically significant improvement in reported quality of life and perceived treatment benefit secondary to overall reported symptom reduction of pain, anxiety, depression, and/or sleeplessness.

### **Secondary Endpoints:** Secondary endpoints consisted of the following:

 Effectiveness: The secondary effectiveness endpoint was overall reduction in median reported symptoms of pain, anxiety, depression, and/or sleeplessness via numeric rating scales at 4, 8, and 12 weeks. This was measured via the following validated tools: Pain intensity and interference- PEG Scale, Anxiety- Generalized Anxiety Disorder 7-item (GAD-7) scale, Depression- Patient Health Questionnaire (PHQ-9), Sleeplessness- PROMIS short form 4a, and overall improvement of quality of life- Patient's Global Impression of Change (PGIC).

The hypothesis-driven criterion was to show that there was a statistically significant reduction in the median reported pain, anxiety, depression, and/or sleeplessness levels of patients using the Nu-V3 device at weeks 4, 8, and 12. The second criterion was intended to show that there was a statistically significant improvement in reported quality of life and perceived treatment benefit secondary to overall reported symptom reduction of pain, anxiety, depression, and/or sleeplessness at weeks 4, 8, and 12.

2. <u>Sub-analyses</u>: The sub-analyses endpoints consisted of the mean number of weeks that pain, anxiety, depression, and sleeplessness response was achieved and sustained, without utilization of another device, during the 8-week intervention. In addition, study sub-analyses included the mean number of weeks to initial benefit from Nu-V3 device use, and the mean medication dosage reduction of short acting pain, anxiolytics, and/or insomnia. The device's



comfort-of-use, and patient's perceived treatment benefit were also captured for sub-analyses.

**Eligibility Criteria Summary:** The study population consisted of both male and female patients, at least 18 years of age.

Key inclusion criteria included the following:

- Participant presents with one or more of the following symptoms: pain, anxiety, depression, and/or sleeplessness
- Participant can commit to follow all protocol study time-points

Key exclusion criteria included the following:

- Participants with a Pacemaker
- Participants with irregular heart rate or a heart rate lower than 60 beats per minute (bradycardia)
- Have had a transplant within the last 2 years
- Have had a heart attack or cardiac bypass surgery within the last 12 months
- History of substance abuse, including prescription drugs, within the last 12 months
- Patients with complaints of dizziness or lightheadedness within the last 3 months
- Women who are pregnant
- Participants with Diabetic Retinopathy
- Current Ear infection
- SBP < 100 and/or DBP < 60
- History of uncontrolled bipolar disorder within the last 12 months
- History of uncontrolled seizures within the last 12 months
- History of Aneurysms
- History of syncope within the last 12 months
- Participants that have had a TIA or stroke within the last 12 months
- Participants with health problems deemed at risk for the study by the Principal Investigator
- Participants with any changes to Pain/Anxiety/Depression/Sleeplessness medications within last 60 days (participants that do not meet this medication change washout period may be delayed until 60-day period is met)
- Participants that are currently under adjudication process for disability support, VA or other

**Accountability:** Patients were exited from the study upon completing the final protocol-required questionnaires. In some cases, patients prematurely exited or withdrew from the study for the following reasons, including but not limited to:

- Not eligible for treatment (including patients who may have signed informed consent and been enrolled).
- Patient experienced a SAE or UPIRTSO.
- Voluntary withdrawal- the patient voluntarily chose not to participate further in the study.



- Lost to follow-up (LTFU) the patient was more than 10 days late to a study visit and
  three documented attempts to contact the patient were unsuccessful. A patient who
  missed a study visit but attended subsequent visit (if required) was no longer considered
  lost to follow-up. A missed visit was considered a protocol deviation and the deviation
  was documented and reported.
- Physician decision in the physician's opinion, it was not in the best interest of the patient to continue study participation.

The tables below summarize patients who exited the study early, as well as those who completed all study participation as per protocol.

| Table 1: Study Exit Summary- Early Exit (<8 weeks) | | | |
|---|---|---|---|
| | Phase I | Phase II | Total Enrolled |
| Voluntary Withdrawal | | | |
| Lost to Follow-Up | | | |
| Physician's Decision | | | |
| SAE / UPIRTSO | | | |
| Other | | | |
| Overall "exited" Patients | | | |

| Table 2: Study Exit Summary (≥ 8 weeks) | | | |
|---|---|---|---|
| | Phase I | Phase II | Total Enrolled |
| Completion of Study as Planned | | | |
| Voluntary Withdrawal | | | |
| Lost to Follow-Up | | | |
| Physician's Decision | | | |
| SAE / UPIRTSO | | | |
| Other | | | |
| Overall "exited" Patients | | | |

Insert Study Exit Analysis Here



## **Section 1.0: Participant Flow**

# ClinicalTrials.gov

A service of the National Institutes of Health

# **Participant Flow Data Preparation Checklist**

Overview: A tabular summary of the participants' progression through each stage of a study by group. Use this checklist with the  $\underline{Participant Flow Template}^{\Delta}$  and  $\underline{Results Data Element Definitions}$ .

| _ | Information to have available for Participant Flow | Term |
|---|---|---|
| | <ul> <li>Conceptual overview of the study design, including the type (e.g., single-group, cross-over, parallel) and any distinct stages (e.g., double-blind then open-label)</li> <li><u>Tip</u>: Have a <u>CONSORT flow diagram</u> available</li> </ul> | Background |
| | <ul> <li>A description of any study events that occurred before participants were<br/>assigned to a study group (e.g., run-in phase, number of screen failures)</li> </ul> | <sup>∆</sup> Pre-assignment<br>Details |
| | <ul> <li>Number of groups that accurately describes the study design from participant assignment to completion. Each group will be reported as a table column.</li> <li><u>Tip</u>: The number of groups is typically equal to the number of unique paths (participant experiences) in a CONSORT flow diagram, from beginning to end.</li> </ul> | Arms/Groups |
| | <ul> <li>For each group, a detailed explanation of the participants and/or interventions</li> <li>Title—A descriptive label for the group (header for the table column). Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1").</li> <li>Description—A detailed explanation of the interventions administered or the groups observed during each stage of the study. Include details about the intervention and the frequency and time period of administration or observation.</li> </ul> | * <sup>A</sup> Arm/Group<br>Title<br><sup>A</sup> Arm/Group<br>Description |
| | Number of distinct stages or intervals of activity in the study | Periods |
| | <ul> <li>If there is more than one stage (Period), each Period will need a unique Title (the default for one Period is "Overall Study").</li> <li>A Period Title should be a descriptive label. For example, "Double-blind (0 to 24 weeks)" and "Open-label (24 to 48 weeks)" are more descriptive than "Period 1" and "Period 2."</li> </ul> | • <sup>∆</sup> Period Title |
| | <ul> <li>For each Period, the number of participants in each group that:</li> <li>Started—Generally, the participants assigned (or randomized) to each group</li> <li>Additional Milestone (optional)—Any important event(s) during study</li> <li>Completed—As defined for the study</li> <li><u>Tip</u>: If the number of participants starting the first Period is different from the total enrolled in the study, explain why in Pre-assignment Details</li> </ul> | • <sup>Δ</sup> Started<br>• <sup>Δ</sup> Completed |
| | <ul> <li>For each Period, the number of participants in each group that dropped out and<br/>the reasons they dropped out</li> </ul> | AReason(s) Not Completed |

\*Required

<sup>∆</sup>Template Field

Edited: 19 August 2014

Figure 1.1- Participant Flow Checklist



#### NU-V3 CONSORT 2010 FLOW DIAGRAM



Figure 1.2- Participant Flow Diagram



| Participant Flor | w Template | Nu-Life Solutions |
|---|---|---|
| Recruitment Detail | s | |
| [*] Pre-assignment | Details | |
| 5 | | |
| Period | | |
| | Phase I | Initial Clinical Study 50 - 100 participants |
| | *Arm/Group Title | |
| *Arm/G | roup Description | |
| | | Number of Participants |
| | *Started | |
| [*] Milestone Title | | |
| [*] Milestone Title | | |
| [*] Milestone Title | | |
| | *Completed | |
| | Not Completed | (automatically calculated) |
| Reason Not Comp | | |
| | luntary Withdrawal | |
| | o Follow-Up (LTFU) | |
| | nysician's Decision | |
| 11 | [*] SAE/ UPIRTSO | |
| [*1 | Protocol Violation | |
| [*] Other | FIOLOCOI VIOIALIOII | |
| []Other | | |
| | Phase II | Expanded Clinical Study 100-200 participants |
| | *Arm/Group Title | |
| *Arm/G | roup Description | |
| | · | Number of Participants |
| | *Started | · |
| [*] Milestone Title | | |
| [*] Milestone Title | | |
| [*] Milestone Title | | |
| | *Completed | |
| | Not Completed | (automatically calculated) |
| Reason Not Comp | • | (automatically catedates) |
| | luntary Withdrawal | |
| | o Follow-Up (LTFU) | |
| | nysician's Decision | |
| []., | [*] SAE/ UPIRTSO | |
| [*1 | Protocol Violation | |
| [*] Other | | |
| *required | | <br>[*] conditionally required |

Figure 1.3- Participant Flow Template



Insert Data Collection Summary Here



### **Section 2.0: Baseline Characteristics**

**Demographics:** The total population consistsed of \_\_\_\_\_ patients. Information on the enrolled patients (n=) patients is provided in the following tables.

# ClinicalTrials.gov

A service of the National Institutes of Health

# **Baseline Characteristics Data Preparation Checklist**

Overview: A tabular summary of all characteristics measured at baseline for each group and overall. The table is similar to "Table 1" in a journal article. Use this checklist with the <u>Results Data Element Definitions</u> and the <u>Simple Results Templates</u><sup>4</sup> for <u>Age; Gender; Race, Ethnicity, Region;</u> and <u>Study Specific Measures</u>.

| Information to have available for Baseline Characteristics | Term |
|---|---|
| <ul> <li>Have a list of all baseline characteristics and the corresponding summary-level<br/>data (similar to Table 1 in a journal article). Age and Gender must be provided.</li> </ul> | Background |
| The number of separate groups for which summary data will be provided. Tip: Generally equal to the number of groups/intervention strategies to which participants were assigned (randomized) at the beginning of the study | Arm/Groups |
| <ul> <li>For each group: <ul> <li>Title—A descriptive label for the group (header for table column). Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1").</li> <li>Description—A detailed explanation of the participants included in the group and the interventions received. This may include a description of how groups of participants were recombined for analysis purposes.</li> </ul> </li> </ul> | *^Arm/Group Title ^Arm/Group Description |
| <ul> <li>Number of participants, in each group and in the entire study population<br/>(total), from whom data were collected and summarized. Participants should<br/>only be represented in one group and in the total (i.e., do not double-count).</li> </ul> | *^Overall Number<br>Baseline Participants |
| <ul> <li>An explanation of the criteria used to determine which participants were<br/>included in the analysis</li> </ul> | Baseline Analysis Population Description |
| Information to have available for each Baseline Measure | Term |
| Information to have available for each Baseline Measure Title—Describe specifically what was measured and will be reported as data Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature). If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values. | |
| Title—Describe specifically what was measured and will be reported as data Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature). If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst). | Term • △Baseline Measure Title △Baseline Measure |
| Title—Describe specifically what was measured and will be reported as data Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature). If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values. The method used to summarize baseline data: Central tendency—E.g., mean, median, geometric mean | Term • <sup>∆</sup> Baseline Measure Title <sup>∆</sup> Baseline Measure Description |
| Title—Describe specifically what was measured and will be reported as data Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature). If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values. The method used to summarize baseline data: Central tendency—E.g., mean, median, geometric mean Number—E.g., count (of participants) For a measure of central tendency, specify a measure that represents "the spread" of the summary data (e.g., standard deviation). | Term **^Baseline Measure Title **Baseline Measure Description **^Measure Type |
| <ul> <li>Title—Describe specifically what was measured and will be reported as data</li> <li>Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature).</li> <li>If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values.</li> <li>The method used to summarize baseline data: <ul> <li>Central tendency—E.g., mean, median, geometric mean</li> <li>Number—E.g., count (of participants)</li> </ul> </li> <li>For a measure of central tendency, specify a measure that represents "the spread" of the summary data (e.g., standard deviation).</li> <li>Tip: This is not applicable for a Number (e.g., count of participants)</li> </ul> | Term **^Baseline Measure Title **Baseline Measure Description **^Measure Type **^Measure of Dispersion |

\*Required <sup>∆</sup>Template Field

Edited: 19 August 2014

Figure 2.1- Baseline Characteristics Checklist



| Baseline Characteristic | Age* | | Nu-Life | e Solutio | ns | |
|---|---|---|---|---|---|---|
| | Group Title | Phase I | Phase II | | Tota | als |
| | Group Description | | | | | |
| Overall Number of B | aseline Participants | | | | | |
| (*) Baseline Analysis Po | oulation Description | | -1 | | | |
| Ana Catanonical | | | | | | |
| Age, Categorical | 19 24 years old | | | 1 | | |
| | 18-24 years old<br>25-34 years old | | | | | |
| | 35-44 years old | | | | | |
| | 45-54 years old | | | | | |
| | 55-64 years old | | | | | |
| | 65-74 years old | | | | | |
| | 75 years or older | | | | | |
| *Unit of Measure | Participants | | | | | |
| | · a | | | | | |
| Age, Customized | | | | | | |
| *Measure Type | *Measure of<br>Dispersion | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One)<br>Not Applicable<br>Standard Deviation<br>Inter-Quartile Range<br>Full Range | | | | | |
| [*] Row/Category Title | | | | | | |
| *Unit of Measure | | | | | | |

<sup>\*</sup>Required

Table 2.2- Baseline Characteristics Template- Age

<sup>[\*]</sup> Conditionally required



# Insert Graphs for Age Distribution Here (examples)





φ Figure 2.3 Distribution of Age Pie Graph





φ Figure 2.4 Distribution of Age Bar Graph

Insert Age Dispersion Statistical Analysis



| Baseline Characteristic | s Template | Sex/Ge | nder at E | Birth* (cl | noose one | e) Nu | ı-Life Sol | utions |
|---|---|---|---|---|---|---|---|---|
| | Grou | p Title | Phase I | | Phase II | | Tot | tals |
| | Group Desc | ription | | | | | | |
| Overall Numbe | r of Baseline Partic | ipants | | | | | | |
| (*) Baseline Analys | (*) Baseline Analysis Population Description | | | | | | | |
| Sex/Gender at Birth: Male, F | emale, Other, Choose | not to a | nswer | | | | | |
| | | Male | | | | | | |
| | I | Female | | | | | | |
| | | Other | | | | | | |
| | Choose not to | answer | | | | | | |
| *Unit of Measure | Participants | | | | | | | |
| Sex/Gender, Customized | | | | | | | | |
| *Measure Type | *Measure of Dispe | rsion | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One)<br>Not Applicable<br>Standard Deviati<br>Inter-Quartile Ran<br>Full Range | on | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| *Unit of Measure | | | | | | | | |

<sup>\*</sup>Required [\*] Conditionally required

Figure 2.5- Baseline Characteristics Template- Sex / Gender



Insert Graphs for Sex / Gender Here (examples)

# **Distribution of Gender**



φ Figure 2.6 Distribution of Gender Pie Graph

### Gender Distribution



φ Figure 2.7 Distribution of Gender Bar Graph

Insert Gender Dispersion Statistical Analysis



| Baseline Characte | eristics Template | Marital Status | * (use at least one) | Nu-Life Solutions |
|---|---|---|---|---|
| | Group Title | Phase I | Phase II | Totals |
| | Group Description | | | |
| | umber of Baseline | | | |
| (t) D II A | Participants | | | |
| (*) Baseline Ar | nalysis Population Description | | | |
| Marital Status: Single, | Married Diversed W | lidowod | | |
| Waritai Status. Siligie, | Single | laowea | | |
| | Married | | | |
| | Divorced | | | |
| | Widowed | | | |
| *Unit of Measure | Participants | | | |
| Offit of Measure | ranticipants | | | |
| Marital Status, Custon | nized | | | |
| *Measure Type | *Measure of<br>Dispersion | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One)<br>Not Applicable<br>Standard Deviation<br>Inter-Quartile Range<br>Full Range | | | |
| [*] Row/Category<br>Title | | | | |
| [*] Row/Category<br>Title | | | | |
| [*] Row/Category<br>Title | | | | |
| *Unit of Measure | | | | |

\*Required

[\*] Conditionally required

Figure 2.8- Baseline Characteristics Template- Marital Status



Insert Graphs for Marital Status Here (examples)

# Marital Status Distribution



φ Figure 2.9 Distribution of Marital Status Bar Graph

# **Marital Status Distribution**



φ Figure 2.10 Distribution of Marital Status Pie Graph

Insert Marital Status Dispersion Statistical Analysis



| Baseline Characteristic | s Template | Primary Language | * (use at lea | st one) | Nu-Life So | olutions |
|---|---|---|---|---|---|---|
| | Group Title | Phase I | Phase II | | Tot | als |
| Gro | up Description | | | | | |
| | per of Baseline | | | | | |
| | Participants | | | | | |
| (*) Baseline Analy | sis Population Description | | | | | |
| B | | | | | , , | |
| Primary Language: Arabic, E<br>Russian, Spanish, Other | Bengali, English, F | rench, German, Hindi/Urdi | u, Japanese, N | landarın, Po | rtuguese, P | unjabi, |
| | Arabic | | | | | |
| | Bengali | | | | | |
| | English | | | | | |
| | French | | | | | |
| | German | | | | | |
| | Hindi/Urdu | | | | | |
| | Japanese | | | | | |
| | Mandarin | | | | | |
| | Portuguese | | | | | |
| | Punjabi | | | | | |
| | Russian | | | | | |
| | Spanish | | | | | |
| | Other | | | | | |
| *Unit of Measure | Participants | | | | | |
| Primary Language, Customi | zed<br>*Measure of | | | | | |
| *Measure Type | Dispersion | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One) Not Applicable Standard Deviation Inter-Quartile Range Full Range | | | | | |
| [*] Row/Category Title | | | | | | |
| [*] Row/Category Title | | | | | | |
| *Unit of Measure | | , | | <u> </u> | | |
| | [*] Conditionally | | | | | |

\*Required [\*] Conditionally required

Figure 2.11- Baseline Characteristics Template- Primary Language



Insert Graphs for Primary Language Here (examples)

# Primary Language Distribution



φ Figure 2.12 Distribution of Primary Language Pie Graph



 $_{
m Figure~2.13~Distribution~of~Primary~Language~Bar~Graph}$ 

Insert Primary Language Dispersion Statistical Analysis Here



| Baseline Characteristic | s Template | Race/E | thnicity* | (use at | least one) | Nu- | Life Solu | tions |
|---|---|---|---|---|---|---|---|---|
| | G | roup Title | Phase I | | Phase II | | To | tals |
| | Group Description | | | | | | | |
| Overall Numbe | r of Baseline Pa | rticipants | | | | | | |
| (*) Baseline Analysi | s Population De | escription | | | | | | |
| Race/Ethnicity: American In<br>Mexican-America/Chicano, F | | | | | | ian, Black/ | African-An | nerican, |
| | Amer | ican Indian | | | | | | |
| Asian-Ameri | can/Oriental/Paci | fic Islander | | | | | | |
| | Asian | East Indian | | | | | | |
| | Black/Africar | n-American | | | | | | |
| | Mexican-Ameri | ca/Chicano | | | | | | |
| | | uerto-Rican | | | | | | |
| | | er Hispanic | | | | | | |
| | White | /Caucasian | | | | | | |
| *Unit of Measure | Doutioinanto | Other | | | | | | |
| Offit of Measure | Participants | | | | | | | |
| Race/Ethnicity, Customized | | | | | | | | |
| *Measure Type | *Measure of D | ispersion | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select O<br>Not Applic<br>Standard De<br>Inter-Quartile<br>Full Ran | able<br>viation<br>Range | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| *Unit of Measure | | | | | | | | |

\*Required

Figure 2.14- Baseline Characteristics Template- Race, Ethnicity

[\*] Conditionally required



### Insert Graphs for Race/Ethnicity Here (examples)



φ Figure 2.15 Distribution of Race/Ethnicity Pie Graph



φ Figure 2.16 Distribution of Race/Ethnicity Bar Graph

Insert Race/Ethnicity Dispersion Statistical Analysis Here



| Baseline Characteristic | s Template | Educatio | n History | /* (use a | at least on | e) N | u-Life Sc | olutions |
|---|---|---|---|---|---|---|---|---|
| | | roup Title | Phase I | | Phase II | | Tot | ale |
| | | Froup Title | riiase i | | riiase ii | | 1 01 | lais |
| Occupation of the section | • | escription | | | | | | |
| Overall Numbe | | <u> </u> | | | | | | |
| (*) Baseline Analys | is Population D | escription | | | | | | |
| Education History: No school<br>graduate- diploma or the eq<br>degree, Bachelor's degree, I | uivalent, Some co | ollege credit- | no degree, | Trade/ted | hnical/voca | ool- no dipl<br>tional train | oma, High<br>ing, Assoc | school<br>iate |
| | No schooling | completed | | | | | | |
| | Nursery school t | o 8th grade | | | | | | |
| S | ome high school, | no diploma | | | | | | |
| High school graduat | te, diploma or the | equivalent | | | | | | |
| Sc | ome college credit | t, no degree | | | | | | |
| Trade/ | technical/vocatio | nal training | | | | | | |
| | Assoc | iate degree | | | | | | |
| | Bache | lor's degree | | | | | | |
| | Mas | ter's degree | | | | | | |
| | Professi | onal degree | | | | | | |
| *Unit of Measure | Participants | | | | | | | |
| Education History, Customiz | zed | | | | | | | |
| *Measure Type | *Measure of D | ispersion | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select C<br>Not Appli<br>Standard De<br>Inter-Quartil<br>Full Rar | cable<br>eviation<br>e Range | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| *Unit of Measure | | | | | | | | |
| *Required | [*] Conditionally | required | | | | | | |

Figure 2.17- Baseline Characteristics Template- Educational History



Insert Graphs for Educational History Measures Here (examples)

## **Education Distribution**



φ Figure 2.18 Distribution of Education Bar Graph

# **Distribution of Education**



P Figure 2.19 Distribution of Education Pie Graph

Insert Education Dispersion Statistical Analysis Here



| Baseline Characteristics Template Service | | Status* ( | use at le | east one) | Nu | -Life Sol | utions | |
|---|---|---|---|---|---|---|---|---|
| | | Froup Title | Phase I | | Phase II | | Tot | als |
| | Group D | escription | | | | | | |
| Overall Numbe | r of Baseline Pa | articipants | | | | | | |
| (*) Baseline Analysi | is Population D | escription | | | | | | |
| Veteran Status: Military Vete | eran, Active Duty | Member, Nev | er Served | in the Arm | ned Forces | | | |
| | Yes, I am a milit | ary veteran | | | | | | |
| Yes, | I am an active du | uty member | | | | | | |
| No, I have neve | er served in the a | rmed forces | | | | | | |
| *Unit of Measure | Participants | | | | | | | |
| First Responder Status: Cur | rent or former Fi | rst Responde | r, Not a Fir | st Respor | ider | | Γ | |
| Yes, I am a curre | ent or former First | t Responder | | | | | | |
| No, I have i | never been a First | t Responder | | | | | | |
| *Unit of Measure | Participants | | | | | | | |
| Service Status, Customized | | | | | | | | |
| *Measure Type | *Measure of D | Dispersion | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select (<br>Not Appli<br>Standard De<br>Inter-Quartil<br>Full Rai | cable<br>eviation<br>e Range | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| *Unit of Measure | | | | | | | | |

\*Required [\*] Conditionally required

Figure 2.20- Baseline Characteristics Template- Service Status



#### Insert Graphs for Service Status Measures Here (examples)



 $\ensuremath{\varphi}$  Figure 2.21 Distribution of Veteran Status Pie Graph

#### **Veteran Status** 140 138 136 Number of Responses 134 132 130 128 126 124 122 120 Active Duty Member Military Veteran No military service Veteran Status

 $\overset{\varphi}{\text{Figure 2.22}}$  Distribution of Veteran Status Bar Graph

### First Responder Status



φ Figure 2.21 Distribution of First Responder Status Pie Graph

### First Responder Status



φ Figure 2.22 Distribution of First Responder Status Bar Graph

Insert Service Status Dispersion Statistical Analysis Here



| Baseline Characteris | tics Template | Stud | dy Specific M | leasure | | Nu-Life | Solutions | |
|---|---|---|---|---|---|---|---|---|
| | Group | Title | Phase I | | Phase II | | Tot | als |
| | Group Descrip | otion | | | | | | |
| Overall Number of | of Baseline Particip | ants | | | | | | |
| (*) Baseline Analysis | Population Descrip | otion | | | | | | |
| [*] Stu | ıdy Specific Measure | Title | | | | | | |
| | Baseline Measure | Title | | | | | | |
| *Measure Type | *Measure of Disper | sion | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One)<br>Not Applicable<br>Standard Deviatio<br>Inter-Quartile Rang<br>Full Range | | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| [*] Row/Category Title | | | | | | | | |
| *Unit of Measure | | | | | | | | |

<sup>\*</sup>Required [\*] Conditionally required

Figure 2.23- Baseline Characteristics Template- Study Specific Measures

Insert Graphs for Study Specific Measures Here (examples)

Insert Study Specific Measures Dispersion Statistical Analysis



### Section 3.0: Outcome Measures and Statistical Analyses

# **Pain**

# **Outcome Measure Data Preparation Checklist**

Overview: A tabular summary of outcome measure results by comparison group. You must report tables for each pre-specified primary and secondary outcome and any appropriate statistical analyses. The outcomes that were pre-specified in the Protocol Section of the record will be available to use and edit during results data entry. You may also include other pre-specified and *post hoc* outcomes. Use this checklist with the <u>Outcome Measure Simple</u>

Results Template and Results Data Element Definitions.

| In | formation to have available for each Outcome Measure | Term |
|---|---|---|
| • | Label the measure as Primary, Secondary, Other Pre-specified, or Post hoc. | • <sup>∆</sup> Outcome Measure<br>Type |
| | Title—Describe specifically what was measured and will be reported as data For example, "Change from baseline in systolic blood pressure at 6 months" specifically describes what was measured and how the outcome data will be reported; "Principle Vital Signs" does not. Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature). For example, a description of how the measure was taken, relevant definitions (e.g., explain "response"), any methods of assessment, and/or calculations that were performed to summarize the data If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst | • <sup>∆</sup> Outcome Measure<br>Title<br><sup>∆</sup> Outcome Measure<br>Description |
| • | possible pain) to allow a reader to properly interpret any reported values. The time point(s) or duration over which a participant was assessed for the measure, and for which data are being reported o For a time-to-event measure—A definition of the stopping rule and the longest duration over which a participant was observed (e.g., from randomization until death, up to 3 years) | • <sup>^</sup> Outcome Measure<br>Time Frame |
| • | The number of separate groups for which summary data will be provided<br><u>Tip</u> : Generally equal to the number of intervention strategies or groups<br>compared | Arm/Groups |
| • | For each group: Title—A descriptive label for the group (header for table column). Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1"). Description—A detailed explanation of the participants included in the group and the interventions received. This may include a description of how groups of participants were recombined for analysis purposes. | • <sup>△</sup> Arm/Group<br>Title<br><sup>△</sup> Arm/Group<br>Description |
| • | Number of participants, in each group, from whom data were collected and summarized. o If the unit of analysis is not participants, also provide the name of the unit (e.g., eyes, lesions) and the number of units [Type/Number Units Analyzed]. | * <sup>A</sup> Number of<br>Participants Analyzed |

\*Required <sup>∆</sup>Template Field



| Information to have available for each Outcome Measure | Term |
|---|---|
| <ul> <li>An explanation of the criteria used to determine which participants were<br/>included in the analysis.</li> </ul> | <sup>∆</sup> Analysis Population<br>Description |
| The method used to summarize outcome data: Central tendency—E.g., mean, median, geometric mean Number—E.g., count, percentage or proportion | • <sup>△</sup> Measure Type |
| <ul> <li>For a measure of central tendency, specify a measure that represents "the spread" of the summary data (e.g., standard deviation) or an estimate of precision (e.g., confidence interval).</li> <li><u>Tip</u>: Either Not applicable or Confidence interval may be appropriate for a Number (e.g., count or percentage of participants).</li> </ul> | * <sup>Δ</sup> Measure of<br>Dispersion/Precision |
| Numerical values for the summary-level data in each group | *Outcome Data |
| <ul> <li>The specific unit associated with the numerical data (e.g., mg/dL)</li> <li>If a proportion or percentage, indicate what it is "of" (e.g., "percentage of participants")</li> </ul> | * <sup>Δ</sup> Unit of Measure |

•Required <sup>∆</sup>Template Field

Figure 3.1- Outcome Measures Checklist- Pain

| Outcome Measure Template | | | | Nu-Life Solutions | | | s |
|---|---|---|---|---|---|---|---|
| * Outcome Measure T | ype (Select One) P | rimary S | Secondary | Other Pre- | specified | Post-Hoc | |
| * Outcome Measure 1 | itle | | | | | | |
| [*] Outcome Measure Descript | tion | | | | | | |
| * Outcome Measure Time Fra | ıme | | | | | | |
| | * Arm / Group Title | Phase I | | Phase II | | То | tal |
| | * Arm / Group Description | Initial 50- | 100 pts | 100-200 pt | ts | 150-300 բ | oatients |
| * Overall Number | er of Participants Analyzed | | | | | | |
| [*] Analy | sis Population Description | | | | | • | |
| *Measure Type | *Measure of Dispersion /<br>Precision | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One) Not Applicable Standard Deviation Standard Error Inter-Quartile Range Full Range% Confidence Interval Geometric Coefficient of Variation | | | | | | |
| [*] Row/Category Title | | | | | | | |
| [*] Row/Category Title | | | | | | | |
| *Unit of Measure | | | ļ. | 1 | | 1 | |

\*Required [\*] Conditionally required

Figure 3.2- Outcome Measures Template- Pain



# **Pain Analysis Graphs**



φ Figure 3.3- Outcome Measures Analysis- Xbar Chart Pain



 $^{\phi}$  Figure 3.4- Outcome Measures Analysis- S Chart Pain

Statistical Analysis Here



#### Outcome Measure - Statistical Analysis (optional)

Overview: The statistical analysis section is a table associated with an Outcome Measure. It summarizes the results of any scientifically appropriate tests of statistical significance or other parameters estimated from the Outcome Measure data. If a statistical analysis is provided, it must include either a P-Value<sup>[\*]</sup> or an Estimation Parameter<sup>[\*]</sup>. You may include as many statistical analyses as is necessary to accommodate all data calculations. Use this checklist with the Results Data Element Definitions.

| | Information to have available for each Statistical Analysis | Term |
|---|---|---|
| | The Outcome Measure group(s) used in the analysis Explain any of the following, if applicable: Null hypothesis for the comparison Power calculation | *Comparison Group Selection<br>Comparison Comments |
| | Was the analysis a test of non-inferiority or equivalence? [Yes or No] If Yes, provide the defined non-inferiority margin. | *Non-inferiority or<br>Equivalence Analysis? [*] Non-inferiority/Equivalence Comments |
| _ | And have one or both of the following: | |
| | <ul> <li>Computed p-value and the statistical method used (e.g., ANOVA, t-test)</li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Adjustments for multiple comparisons or covariates</li> <li>Degrees of freedom</li> <li>A priori threshold for statistical significance (e.g., &lt; 0.05)</li> </ul> </li> </ul> | P-Value and Method |
| | <ul> <li>Value of any parameter derived from the outcome measure data (e.g., hazard ratio, mean difference, correlation coefficient)</li> <li>Any of the following, if available: <ul> <li>Confidence Interval</li> <li>Standard deviation or standard error</li> </ul> </li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Directionality of comparison. For subtraction (i.e., A – B or B – A) or a ratio (i.e., A/B or B/A)</li> </ul> </li> </ul> | Estimation Parameter and Value Confidence Interval Parameter Dispersion Estimation Comments |

\*Required

[\*] Conditionally required

Figure 3.5- Statistical Analysis Checklist- Pain

Insert Summary of Results Here



# **Anxiety**

# **Outcome Measure Data Preparation Checklist**

Overview: A tabular summary of outcome measure results by comparison group. You must report tables for each pre-specified primary and secondary outcome and any appropriate statistical analyses. The outcomes that were pre-specified in the Protocol Section of the record will be available to use and edit during results data entry. You may also include other pre-specified and post hoc outcomes. Use this checklist with the Outcome Measure Simple Results Template A and Results Data Element Definitions.

| In | formation to have available for each Outcome Measure | Term |
|---|---|---|
| • | Label the measure as Primary, Secondary, Other Pre-specified, or Post hoc. | • <sup>∆</sup> Outcome Measure<br>Type |
| • • | Title—Describe specifically what was measured and will be reported as data For example, "Change from baseline in systolic blood pressure at 6 months" specifically describes what was measured and how the outcome data will be reported; "Principle Vital Signs" does not. Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature). For example, a description of how the measure was taken, relevant definitions (e.g., explain "response"), any methods of assessment, and/or calculations that were performed to summarize the data If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values. | • <sup>Δ</sup> Outcome Measure<br>Title<br><sup>Δ</sup> Outcome Measure<br>Description |
| • | The time point(s) or duration over which a participant was assessed for the measure, and for which data are being reported o For a time-to-event measure—A definition of the stopping rule and the longest duration over which a participant was observed (e.g., from randomization until death, up to 3 years) | • <sup>∆</sup> Outcome Measure<br>Time Frame |
| • • | The number of separate groups for which summary data will be provided<br><u>Tip</u> : Generally equal to the number of intervention strategies or groups<br>compared | Arm/Groups |
| • | For each group: Title—A descriptive label for the group (header for table column). Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1"). Description—A detailed explanation of the participants included in the group and the interventions received. This may include a description of how groups of participants were recombined for analysis purposes. | * <sup>Δ</sup> Arm/Group<br>Title<br><sup>Δ</sup> Arm/Group<br>Description |
| • | Number of participants, in each group, from whom data were collected and summarized. o If the unit of analysis is not participants, also provide the name of the unit (e.g., eyes, lesions) and the number of units [Type/Number Units Analyzed]. | *^Number of<br>Participants Analyzed |

\*Required <sup>A</sup>Template Field



| Information to have available for each Outcome Measure | Term |
|---|---|
| <ul> <li>An explanation of the criteria used to determine which participants were<br/>included in the analysis.</li> </ul> | <sup>∆</sup> Analysis Population<br>Description |
| <ul> <li>The method used to summarize outcome data:</li> <li>Central tendency—E.g., mean, median, geometric mean</li> <li>Number—E.g., count, percentage or proportion</li> </ul> | • <sup>△</sup> Measure Type |
| <ul> <li>For a measure of central tendency, specify a measure that represents "the spread" of the summary data (e.g., standard deviation) or an estimate of precision (e.g., confidence interval).</li> <li>Tip: Either Not applicable or Confidence interval may be appropriate for a Number (e.g., count or percentage of participants).</li> </ul> | * <sup>Δ</sup> Measure of<br>Dispersion/Precision |
| Numerical values for the summary-level data in each group | *Outcome Data |
| <ul> <li>The specific unit associated with the numerical data (e.g., mg/dL)</li> <li>If a proportion or percentage, indicate what it is "of" (e.g., "percentage of participants")</li> </ul> | • <sup>∆</sup> Unit of Measure |

^Template Field

Figure 3.6- Outcome Measures Checklist- Anxiety

| Outcome Measure Template | | | | Nu-Life Solutions | | | ıs |
|---|---|---|---|---|---|---|---|
| * Outcome Measure T | ype (Select One) P | elect One) Primary Secondary | | Other Pre-specified | | Post-Hoc | |
| * Outcome Measure T | itle | | | | | | |
| [*] Outcome Measure Descript | ion | | | | | | |
| * Outcome Measure Time Fra | me | | | | | | |
| | * Arm / Group Title | Phase I | | Phase II | | То | tal |
| | * Arm / Group Description | Initial 50- | 100 pts | 100-200 p | ts | 150-300 բ | oatients |
| * Overall Number | er of Participants Analyzed | | | | | | |
| [*] Analy | [*] Analysis Population Description | | | | | | |
| *Measure Type | *Measure of Dispersion /<br>Precision | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One) Not Applicable Standard Deviation Standard Error Inter-Quartile Range Full Range% Confidence Interval Geometric Coefficient of Variation | | | | | | |
| [*] Row/Category Title | | | | | | | |
| [*] Row/Category Title | | | | | | | |
| *Unit of Measure | | | | | | | |

\*Required [\*] Conditionally required

Figure 3.7- Outcome Measures Template- Anxiety



# Insert Anxiety Analysis Graphs Here



φ Figure 3.8- Outcome Measures Analysis- Xbar Chart Anxiety



φ Figure 3.9- Outcome Measures Analysis- S Chart Anxiety

Statistical Analysis Here



#### Outcome Measure - Statistical Analysis (optional)

Overview: The statistical analysis section is a table associated with an Outcome Measure. It summarizes the results of any scientifically appropriate tests of statistical significance or other parameters estimated from the Outcome Measure data. If a statistical analysis is provided, it must include either a P-Value<sup>[\*]</sup> or an Estimation Parameter<sup>[\*]</sup>. You may include as many statistical analyses as is necessary to accommodate all data calculations. Use this checklist with the Results Data Element Definitions.

| | Information to have available for each Statistical Analysis | Term |
|---|---|---|
| | The Outcome Measure group(s) used in the analysis Explain any of the following, if applicable: Null hypothesis for the comparison Power calculation | *Comparison Group Selection<br>Comparison Comments |
| | Was the analysis a test of non-inferiority or equivalence? [Yes or No] If Yes, provide the defined non-inferiority margin. | *Non-inferiority or<br>Equivalence Analysis? [*] Non-inferiority/Equivalence Comments |
| _ | And have one or both of the following: | |
| | <ul> <li>Computed p-value and the statistical method used (e.g., ANOVA, t-test)</li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Adjustments for multiple comparisons or covariates</li> <li>Degrees of freedom</li> <li>A priori threshold for statistical significance (e.g., &lt; 0.05)</li> </ul> </li> </ul> | P-Value and Method |
| | <ul> <li>Value of any parameter derived from the outcome measure data (e.g., hazard ratio, mean difference, correlation coefficient)</li> <li>Any of the following, if available: <ul> <li>Confidence Interval</li> <li>Standard deviation or standard error</li> </ul> </li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Directionality of comparison. For subtraction (i.e., A – B or B – A) or a ratio (i.e., A/B or B/A)</li> </ul> </li> </ul> | Estimation Parameter and Value Confidence Interval Parameter Dispersion Estimation Comments |

\*Required

[\*] Conditionally required

Figure 3.10- Statistical Analysis Checklist- Anxiety

Insert Summary of Results Here



#### **Depression**

# **Outcome Measure Data Preparation Checklist**

Overview: A tabular summary of outcome measure results by comparison group. You must report tables for each pre-specified primary and secondary outcome and any appropriate statistical analyses. The outcomes that were pre-specified in the Protocol Section of the record will be available to use and edit during results data entry. You may also include other pre-specified and post hoc outcomes. Use this checklist with the Outcome Measure Simple Results Template A and Results Data Element Definitions.

| Information to have available for each Outcome Measure | Term |
|---|---|
| Label the measure as Primary, Secondary, Other Pre-specified, or Post hoc. | * <sup>∆</sup> Outcome Measure<br>Type |
| <ul> <li>Title—Describe specifically what was measured and will be reported as data <ul> <li>For example, "Change from baseline in systolic blood pressure at 6 months" specifically describes what was measured and how the outcome data will be reported; "Principle Vital Signs" does not.</li> </ul> </li> <li>Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature).</li> <li>For example, a description of how the measure was taken, relevant definitions (e.g., explain "response"), any methods of assessment, and/or calculations that were performed to summarize the data</li> <li>If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values.</li> </ul> | * <sup>Δ</sup> Outcome Measure<br>Title<br><sup>Δ</sup> Outcome Measure<br>Description |
| The time point(s) or duration over which a participant was assessed for the measure, and for which data are being reported For a time-to-event measure—A definition of the stopping rule and the longest duration over which a participant was observed (e.g., from randomization until death, up to 3 years) | * <sup>^</sup> Outcome Measure<br>Time Frame |
| The number of separate groups for which summary data will be provided <u>Tip</u> : Generally equal to the number of intervention strategies or groups compared | Arm/Groups |
| <ul> <li>For each group: <ul> <li>Title—A descriptive label for the group (header for table column). Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1").</li> <li>Description—A detailed explanation of the participants included in the group and the interventions received. This may include a description of how groups of participants were recombined for analysis purposes.</li> </ul> </li> </ul> | •^Arm/Group<br>Title<br>^Arm/Group<br>Description |
| <ul> <li>Number of participants, in each group, from whom data were collected and summarized.</li> <li>If the unit of analysis is not participants, also provide the name of the unit (e.g., eyes, lesions) and the number of units [Type/Number Units Analyzed].</li> </ul> | * <sup>∆</sup> Number of<br>Participants Analyzed |

\*Required <sup>∆</sup>Template Field



| Information to have available for each Outcome Measure | Term |
|---|---|
| <ul> <li>An explanation of the criteria used to determine which participants were<br/>included in the analysis.</li> </ul> | <sup>∆</sup> Analysis Population<br>Description |
| The method used to summarize outcome data: Central tendency—E.g., mean, median, geometric mean Number—E.g., count, percentage or proportion | • <sup>∆</sup> Measure Type |
| <ul> <li>For a measure of central tendency, specify a measure that represents "the spread" of the summary data (e.g., standard deviation) or an estimate of precision (e.g., confidence interval).</li> <li>Tip: Either Not applicable or Confidence interval may be appropriate for a Number (e.g., count or percentage of participants).</li> </ul> | * <sup>A</sup> Measure of<br>Dispersion/Precision |
| Numerical values for the summary-level data in each group | *Outcome Data |
| <ul> <li>The specific unit associated with the numerical data (e.g., mg/dL)</li> <li>If a proportion or percentage, indicate what it is "of" (e.g., "percentage of participants")</li> </ul> | • <sup>∆</sup> Unit of Measure |
| | *Required |

\*Required ∆Template Field

Figure 3.11- Outcome Measures Checklist- Depression

| Outcome Measure Template De | | | epression | | | Nu-Life Solutions | |
|---|---|---|---|---|---|---|---|
| * Outcome Measure T | ype (Select One) | Primary | Secondary | Other Pre-specified | | Post-Hoc | |
| * Outcome Measure T | itle | | | | | | |
| [*] Outcome Measure Descript | ion | | | | | | |
| * Outcome Measure Time Fra | ime | | | | | | |
| * Arm / Group Title | | | Phase I | | Phase II | | Total |
| * Arm / Group Description | | | Initial 50-100 pts | | 100-200 pts | | 150-300 patients |
| * Overall Number of Participants Analyzed | | | | | | | |
| [*] Analysis Population Description | | | | • | | - | |
| *Measure Type | *Measure of Dispersion<br>Precision | 1 | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One) Not Applicable Standard Deviation Standard Error Inter-Quartile Range Full Range% Confidence Interval Geometric Coefficient o | f | | | | | |
| [*] Row/Category Title | | | | | | | |
| [*] Row/Category Title | | | | | | | |
| *Unit of Measure | | | , | + | 1 | , | |

\*Required [\*] Conditionally required

Figure 3.12- Outcome Measures Template- Depression


# Insert Depression Analysis Graphs Here



φ Figure 3.13- Outcome Measures Analysis- Xbar Chart Depression



φ Figure 3.14- Outcome Measures Analysis- S Chart Depression

Statistical Analysis Here



Overview: The statistical analysis section is a table associated with an Outcome Measure. It summarizes the results of any scientifically appropriate tests of statistical significance or other parameters estimated from the Outcome Measure data. If a statistical analysis is provided, it must include either a P-Value<sup>[\*]</sup> or an Estimation Parameter<sup>[\*]</sup>. You may include as many statistical analyses as is necessary to accommodate all data calculations. Use this checklist with the Results Data Element Definitions.

| | Information to have available for each Statistical Analysis | Term |
|---|---|---|
| | The Outcome Measure group(s) used in the analysis Explain any of the following, if applicable: Null hypothesis for the comparison Power calculation | *Comparison Group Selection<br>Comparison Comments |
| | Was the analysis a test of non-inferiority or equivalence? [Yes or No] If Yes, provide the defined non-inferiority margin. | *Non-inferiority or<br>Equivalence Analysis? [*] Non-inferiority/Equivalence Comments |
| _ | And have one or both of the following: | |
| | <ul> <li>Computed p-value and the statistical method used (e.g., ANOVA, t-test)</li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Adjustments for multiple comparisons or covariates</li> <li>Degrees of freedom</li> <li>A priori threshold for statistical significance (e.g., &lt; 0.05)</li> </ul> </li> </ul> | P-Value and Method |
| | <ul> <li>Value of any parameter derived from the outcome measure data (e.g., hazard ratio, mean difference, correlation coefficient)</li> <li>Any of the following, if available: <ul> <li>Confidence Interval</li> <li>Standard deviation or standard error</li> </ul> </li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Directionality of comparison. For subtraction (i.e., A – B or B – A) or a ratio (i.e., A/B or B/A)</li> </ul> </li> </ul> | Estimation Parameter and Value Confidence Interval Parameter Dispersion Estimation Comments |

\*Required

[\*] Conditionally required

Figure 3.15- Statistical Analysis Checklist- Depression

Insert Summary of Results Here



# **Sleeplessness**

# **Outcome Measure Data Preparation Checklist**

Overview: A tabular summary of outcome measure results by comparison group. You must report tables for each pre-specified primary and secondary outcome and any appropriate statistical analyses. The outcomes that were pre-specified in the Protocol Section of the record will be available to use and edit during results data entry. You may also include other pre-specified and post hoc outcomes. Use this checklist with the Outcome Measure Simple Results Template A and Results Data Element Definitions.

| Information to have available for each Outcome Measure | Term |
|---|---|
| Label the measure as Primary, Secondary, Other Pre-specified, or Post hoc. | •^Outcome Measure<br>Type |
| <ul> <li>Title—Describe specifically what was measured and will be reported as data</li> <li>For example, "Change from baseline in systolic blood pressure at 6 months" specifically describes what was measured and how the outcome data will be reported; "Principle Vital Signs" does not.</li> <li>Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature).</li> <li>For example, a description of how the measure was taken, relevant definitions (e.g., explain "response"), any methods of assessment, and/or calculations that were performed to summarize the data</li> <li>If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values.</li> </ul> | • <sup>∆</sup> Outcome Measure<br>Title<br><sup>∆</sup> Outcome Measure<br>Description |
| <ul> <li>The time point(s) or duration over which a participant was assessed for the measure, and for which data are being reported</li> <li>For a time-to-event measure—A definition of the stopping rule and the longest duration over which a participant was observed (e.g., from randomization until death, up to 3 years)</li> </ul> | • <sup>△</sup> Outcome Measure<br>Time Frame |
| <ul> <li>The number of separate groups for which summary data will be provided</li> <li><u>Tip</u>: Generally equal to the number of intervention strategies or groups compared</li> </ul> | Arm/Groups |
| <ul> <li>For each group: <ul> <li>Title—A descriptive label for the group (header for table column). Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1").</li> <li>Description—A detailed explanation of the participants included in the group and the interventions received. This may include a description of how groups of participants were recombined for analysis purposes.</li> </ul> </li> </ul> | • <sup>∆</sup> Arm/Group<br>Title<br><sup>△</sup> Arm/Group<br>Description |
| <ul> <li>Number of participants, in each group, from whom data were collected and summarized.</li> <li>If the unit of analysis is not participants, also provide the name of the unit (e.g., eyes, lesions) and the number of units [Type/Number Units Analyzed].</li> </ul> | *^Number of<br>Participants Analyzed |

\*Required <sup>A</sup>Template Field



| Information to have available for each Outcome Measure | Term |
|---|---|
| <ul> <li>An explanation of the criteria used to determine which participants were<br/>included in the analysis.</li> </ul> | <sup>∆</sup> Analysis Population<br>Description |
| The method used to summarize outcome data: Central tendency—E.g., mean, median, geometric mean Number—E.g., count, percentage or proportion | • <sup>∆</sup> Measure Type |
| <ul> <li>For a measure of central tendency, specify a measure that represents "the spread" of the summary data (e.g., standard deviation) or an estimate of precision (e.g., confidence interval).</li> <li><u>Tip</u>: Either Not applicable or Confidence interval may be appropriate for a Number (e.g., count or percentage of participants).</li> </ul> | * <sup>Δ</sup> Measure of<br>Dispersion/Precision |
| Numerical values for the summary-level data in each group | *Outcome Data |
| <ul> <li>The specific unit associated with the numerical data (e.g., mg/dL)</li> <li>If a proportion or percentage, indicate what it is "of" (e.g., "percentage of participants")</li> </ul> | • <sup>∆</sup> Unit of Measure |

<sup>∆</sup>Template Field

Figure 3.16- Outcome Measures Checklist- Sleeplessness

| Outcome Measure Tem | eplessne | ss | | Nu-Life | Solution | ıs | |
|---|---|---|---|---|---|---|---|
| * Outcome Measure T | ype (Select One) Pr | imary S | econdary | Other Pre- | specified | Post-Hoc | |
| * Outcome Measure 1 | Title Title | | | | | | |
| [*] Outcome Measure Descrip | tion | | | | | | |
| * Outcome Measure Time Fra | ame | | | | | | |
| | * Arm / Group Title | Phase I | | Phase II | | To | tal |
| | * Arm / Group Description | Initial 50-1 | 00 pts | 100-200 pt | s | 150-300 | oatients |
| * Overall Number | er of Participants Analyzed | | | | | | |
| [*] Analy | | | 1 | | • | | |
| *Measure Type | *Measure of Dispersion /<br>Precision | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One) Not Applicable Standard Deviation Standard Error Inter-Quartile Range Full Range% Confidence Interval Geometric Coefficient of Variation | | | | | | |
| [*] Row/Category Title | | | | | | | |
| [*] Row/Category Title | | | | | | | |
| *Unit of Measure | | | | 1 | | 1 | |

[\*] Conditionally required \*Required

Figure 3.17- Outcome Measures Template- Sleeplessness



# Insert Sleeplessness Analysis Graphs Here



Figure 3.18- Outcome Measures Analysis- Xbar Chart Sleeplessness



φ Figure 3.19- Outcome Measures Analysis- S Chart Sleeplessness

Statistical Analysis Here



Overview: The statistical analysis section is a table associated with an Outcome Measure. It summarizes the results of any scientifically appropriate tests of statistical significance or other parameters estimated from the Outcome Measure data. If a statistical analysis is provided, it must include either a P-Value<sup>[\*]</sup> or an Estimation Parameter<sup>[\*]</sup>. You may include as many statistical analyses as is necessary to accommodate all data calculations. Use this checklist with the Results Data Element Definitions.

| | Information to have available for each Statistical Analysis | Term |
|---|---|---|
| | The Outcome Measure group(s) used in the analysis Explain any of the following, if applicable: Null hypothesis for the comparison Power calculation | *Comparison Group Selection<br>Comparison Comments |
| | Was the analysis a test of non-inferiority or equivalence? [Yes or No] If Yes, provide the defined non-inferiority margin. | *Non-inferiority or<br>Equivalence Analysis? [*] Non-inferiority/Equivalence Comments |
| _ | And have one or both of the following: | |
| | <ul> <li>Computed p-value and the statistical method used (e.g., ANOVA, t-test)</li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Adjustments for multiple comparisons or covariates</li> <li>Degrees of freedom</li> <li>A priori threshold for statistical significance (e.g., &lt; 0.05)</li> </ul> </li> </ul> | P-Value and Method |
| | <ul> <li>Value of any parameter derived from the outcome measure data (e.g., hazard ratio, mean difference, correlation coefficient)</li> <li>Any of the following, if available: <ul> <li>Confidence Interval</li> <li>Standard deviation or standard error</li> </ul> </li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Directionality of comparison. For subtraction (i.e., A – B or B – A) or a ratio (i.e., A/B or B/A)</li> </ul> </li> </ul> | Estimation Parameter and Value Confidence Interval Parameter Dispersion Estimation Comments |

\*Required

[\*] Conditionally required

Figure 3.20- Statistical Analysis Checklist- Sleeplessness

Insert Summary of Results Here



# **Quality of Life**

# **Outcome Measure Data Preparation Checklist**

Overview: A tabular summary of outcome measure results by comparison group. You must report tables for each pre-specified primary and secondary outcome and any appropriate statistical analyses. The outcomes that were pre-specified in the Protocol Section of the record will be available to use and edit during results data entry. You may also include other pre-specified and post hoc outcomes. Use this checklist with the Outcome Measure Simple Results Template A and Results Data Element Definitions.

| ln | formation to have available for each Outcome Measure | Term |
|---|---|---|
| • | Label the measure as Primary, Secondary, Other Pre-specified, or Post hoc. | • <sup>∆</sup> Outcome Measure<br>Type |
| • | Title—Describe specifically what was measured and will be reported as data For example, "Change from baseline in systolic blood pressure at 6 months" specifically describes what was measured and how the outcome data will be reported; "Principle Vital Signs" does not. Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature). For example, a description of how the measure was taken, relevant definitions (e.g., explain "response"), any methods of assessment, and/or calculations that were performed to summarize the data If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values. | • <sup>Δ</sup> Outcome Measure<br>Title<br><sup>Δ</sup> Outcome Measure<br>Description |
| • | The time point(s) or duration over which a participant was assessed for the measure, and for which data are being reported o For a time-to-event measure—A definition of the stopping rule and the longest duration over which a participant was observed (e.g., from randomization until death, up to 3 years) | • <sup>∆</sup> Outcome Measure<br>Time Frame |
| • • | The number of separate groups for which summary data will be provided<br><u>Tip</u> : Generally equal to the number of intervention strategies or groups<br>compared | Arm/Groups |
| • | For each group: Title—A descriptive label for the group (header for table column). Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1"). Description—A detailed explanation of the participants included in the group and the interventions received. This may include a description of how groups of participants were recombined for analysis purposes. | • <sup>∆</sup> Arm/Group<br>Title<br><sup>∆</sup> Arm/Group<br>Description |
| • | Number of participants, in each group, from whom data were collected and summarized. o If the unit of analysis is not participants, also provide the name of the unit (e.g., eyes, lesions) and the number of units [Type/Number Units Analyzed]. | * <sup>4</sup> Number of<br>Participants Analyzed |

\*Required <sup>^</sup>Template Field



| Information to have available for each Outcome Measure | Term |
|---|---|
| <ul> <li>An explanation of the criteria used to determine which participants were<br/>included in the analysis.</li> </ul> | <sup>∆</sup> Analysis Population<br>Description |
| The method used to summarize outcome data: Central tendency—E.g., mean, median, geometric mean Number—E.g., count, percentage or proportion | • <sup>△</sup> Measure Type |
| <ul> <li>For a measure of central tendency, specify a measure that represents "the spread" of the summary data (e.g., standard deviation) or an estimate of precision (e.g., confidence interval).</li> <li>Tip: Either Not applicable or Confidence interval may be appropriate for a Number (e.g., count or percentage of participants).</li> </ul> | * <sup>A</sup> Measure of<br>Dispersion/Precision |
| Numerical values for the summary-level data in each group | *Outcome Data |
| <ul> <li>The specific unit associated with the numerical data (e.g., mg/dL)</li> <li>If a proportion or percentage, indicate what it is "of" (e.g., "percentage of participants")</li> </ul> | * <sup>Δ</sup> Unit of Measure |

\*Required ∆Template Field

Figure 3.21- Outcome Measures Checklist- QOL

| Outcome Measure Tem | y of Life- | PGIC | | Nu-Life | Solution | ıs | |
|---|---|---|---|---|---|---|---|
| * Outcome Measure T | ype (Select One) Pr | rimary S | Secondary | Other Pre- | specified | Post-Hoc | |
| * Outcome Measure 1 | itle | | | | | | |
| [*] Outcome Measure Descript | ion | | | | | | |
| * Outcome Measure Time Fra | me | | | | | | |
| | * Arm / Group Title | Phase I | | Phase II | | To | tal |
| | * Arm / Group Description | Initial 50- | 100 pts | 100-200 pt | ts | 150-300 | oatients |
| * Overall Number | er of Participants Analyzed | | | | | | |
| [*] Analy | [*] Analysis Population Description | | | • | | • | |
| *Measure Type | *Measure of Dispersion /<br>Precision | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One) Not Applicable Standard Deviation Standard Error Inter-Quartile Range Full Range% Confidence Interval Geometric Coefficient of Variation | | | | | | |
| [*] Row/Category Title | | | | | | | |
| [*] Row/Category Title | | | | | | | |
| *Unit of Measure | | | | | | • | |

\*Required [\*] Conditionally required

Figure 3.22- Outcome Measures Template- Quality of Life



# Insert Quality of Life Analysis Graphs Here



Figure 3.23- Outcome Measures Analysis- Xbar Chart QOL Level



Figure 3.24- Outcome Measures Analysis- S Chart QOL Level

Statistical Analysis Here



Overview: The statistical analysis section is a table associated with an Outcome Measure. It summarizes the results of any scientifically appropriate tests of statistical significance or other parameters estimated from the Outcome Measure data. If a statistical analysis is provided, it must include either a P-Value<sup>[\*]</sup> or an Estimation Parameter<sup>[\*]</sup>. You may include as many statistical analyses as is necessary to accommodate all data calculations. Use this checklist with the Results Data Element Definitions.

| | Information to have available for each Statistical Analysis | Term |
|---|---|---|
| | The Outcome Measure group(s) used in the analysis Explain any of the following, if applicable: Null hypothesis for the comparison Power calculation | *Comparison Group Selection<br>Comparison Comments |
| | Was the analysis a test of non-inferiority or equivalence? [Yes or No] If Yes, provide the defined non-inferiority margin. | *Non-inferiority or<br>Equivalence Analysis? [*] Non-inferiority/Equivalence Comments |
| _ | And have one or both of the following: | |
| | <ul> <li>Computed p-value and the statistical method used (e.g., ANOVA, t-test)</li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Adjustments for multiple comparisons or covariates</li> <li>Degrees of freedom</li> <li>A priori threshold for statistical significance (e.g., &lt; 0.05)</li> </ul> </li> </ul> | P-Value and Method |
| | <ul> <li>Value of any parameter derived from the outcome measure data (e.g., hazard ratio, mean difference, correlation coefficient)</li> <li>Any of the following, if available: <ul> <li>Confidence Interval</li> <li>Standard deviation or standard error</li> </ul> </li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Directionality of comparison. For subtraction (i.e., A – B or B – A) or a ratio (i.e., A/B or B/A)</li> </ul> </li> </ul> | Estimation Parameter and Value Confidence Interval Parameter Dispersion Estimation Comments |

\*Required

[\*] Conditionally required

Figure 3.25- Statistical Analysis Checklist- Quality of Life Level

Insert Summary of Results Here



# Reduction of Total Daily Dosage: Indication- Relevant Medications Taken (Baseline, 30, 60, 90 Days)

# **Outcome Measure Data Preparation Checklist**

Overview: A tabular summary of outcome measure results by comparison group. You must report tables for each pre-specified primary and secondary outcome and any appropriate statistical analyses. The outcomes that were pre-specified in the Protocol Section of the record will be available to use and edit during results data entry. You may also include other pre-specified and post hoc outcomes. Use this checklist with the Outcome Measure Simple Results Template A and Results Data Element Definitions.

| Inf | formation to have available for each Outcome Measure | Term |
|---|---|---|
| • | Label the measure as Primary, Secondary, Other Pre-specified, or Post hoc. | • <sup>∆</sup> Outcome Measure<br>Type |
| • | Title—Describe specifically what was measured and will be reported as data For example, "Change from baseline in systolic blood pressure at 6 months" specifically describes what was measured and how the outcome data will be reported; "Principle Vital Signs" does not. Description—Any elaboration needed to understand the measure and the reported data. Information should be written for a public audience (i.e., not specialists in your field, but general readers of the medical literature). For example, a description of how the measure was taken, relevant definitions (e.g., explain "response"), any methods of assessment, and/or calculations that were performed to summarize the data If the measure was based on a scale, explain any numerical categories or provide the range and direction of possible scores (0=no pain; 10=worst possible pain) to allow a reader to properly interpret any reported values. | * <sup>Δ</sup> Outcome Measure<br>Title<br><sup>Δ</sup> Outcome Measure<br>Description |
| • | The time point(s) or duration over which a participant was assessed for the measure, and for which data are being reported o For a time-to-event measure—A definition of the stopping rule and the longest duration over which a participant was observed (e.g., from randomization until death, up to 3 years) | * <sup>A</sup> Outcome Measure<br>Time Frame |
| • • | The number of separate groups for which summary data will be provided<br><u>Tip</u> : Generally equal to the number of intervention strategies or groups<br>compared | Arm/Groups |
| • | For each group: Title—A descriptive label for the group (header for table column). Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1"). Description—A detailed explanation of the participants included in the group and the interventions received. This may include a description of how groups of participants were recombined for analysis purposes. | * <sup>Δ</sup> Arm/Group<br>Title<br><sup>Δ</sup> Arm/Group<br>Description |
| • | Number of participants, in each group, from whom data were collected and summarized. o If the unit of analysis is not participants, also provide the name of the unit (e.g., eyes, lesions) and the number of units [Type/Number Units Analyzed]. | • <sup>△</sup> Number of<br>Participants Analyzed |

\*Required <sup>∆</sup>Template Field



| Information to have available for each Outcome Measure | Term |
|---|---|
| <ul> <li>An explanation of the criteria used to determine which participants were<br/>included in the analysis.</li> </ul> | <sup>∆</sup> Analysis Population<br>Description |
| The method used to summarize outcome data: Central tendency—E.g., mean, median, geometric mean Number—E.g., count, percentage or proportion | • <sup>△</sup> Measure Type |
| <ul> <li>For a measure of central tendency, specify a measure that represents "the spread" of the summary data (e.g., standard deviation) or an estimate of precision (e.g., confidence interval).</li> <li>Tip: Either Not applicable or Confidence interval may be appropriate for a Number (e.g., count or percentage of participants).</li> </ul> | * <sup>A</sup> Measure of<br>Dispersion/Precision |
| Numerical values for the summary-level data in each group | *Outcome Data |
| <ul> <li>The specific unit associated with the numerical data (e.g., mg/dL)</li> <li>If a proportion or percentage, indicate what it is "of" (e.g., "percentage of participants")</li> </ul> | * <sup>∆</sup> Unit of Measure |

<sup>∆</sup>Template Field

Figure 3.26- Outcome Measures Checklist- Relevant Medication Dosage Decrease

| Outcome Measure Tem | nt Medic<br>ge Decre | | | Nu-Life | Solution | ıs | |
|---|---|---|---|---|---|---|---|
| * Outcome Measure T | ype (Select One) Pri | imary S | econdary | Other Pre- | -specified | Post-Hoc | |
| * Outcome Measure 1 | itle | | | | | | |
| [*] Outcome Measure Descript | ion | | | | | | |
| * Outcome Measure Time Fra | nme | | | | | | |
| | * Arm / Group Title | Phase I | | Phase II | | То | tal |
| | * Arm / Group Description | Initial 50- | I00 pts | 100-200 pt | ts | 150-300 patients | |
| * Overall Number | er of Participants Analyzed | | | | | | |
| [*] Analy | sis Population Description | | | | | | |
| *Measure Type | *Measure of Dispersion / Precision | | | | | | |
| (Select One) Count of Participants Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units | (Select One) Not Applicable Standard Deviation Standard Error Inter-Quartile Range Full Range% Confidence Interval Geometric Coefficient of Variation | | | | | | |
| [*] Row/Category Title | | | | | | | |
| [*] Row/Category Title<br>*Unit of Measure | | | | | | | |

\*Required [\*] Conditionally required

Figure 3.27- Outcome Measures Template- Relevant Medication Dosage Decrease



Insert Relevant Medication Dosage Decrease Analysis Graphs Here



Ψ Figure 3.28- Outcome Measures Analysis- Xbar Chart Relevant Medication Dosage Decrease



φ Figure 3.29- Outcome Measures Analysis- S Chart Relevant Medication Dosage Decrease

Insert Relevant Medication Dosage Decrease Statistical Analysis Here



Overview: The statistical analysis section is a table associated with an Outcome Measure. It summarizes the results of any scientifically appropriate tests of statistical significance or other parameters estimated from the Outcome Measure data. If a statistical analysis is provided, it must include either a P-Value<sup>[\*]</sup> or an Estimation Parameter<sup>[\*]</sup>. You may include as many statistical analyses as is necessary to accommodate all data calculations. Use this checklist with the Results Data Element Definitions.

| | Information to have available for each Statistical Analysis | Term |
|---|---|---|
| | The Outcome Measure group(s) used in the analysis Explain any of the following, if applicable: Null hypothesis for the comparison Power calculation | *Comparison Group Selection<br>Comparison Comments |
| | Was the analysis a test of non-inferiority or equivalence? [Yes or No] If Yes, provide the defined non-inferiority margin. | *Non-inferiority or<br>Equivalence Analysis?<br><sup>(*)</sup> Non-inferiority/Equivalence<br>Comments |
| _ | And have one or both of the following: | |
| | <ul> <li>Computed p-value and the statistical method used (e.g., ANOVA, t-test)</li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Adjustments for multiple comparisons or covariates</li> <li>Degrees of freedom</li> <li>A priori threshold for statistical significance (e.g., &lt; 0.05)</li> </ul> </li> </ul> | P-Value and Method |
| | <ul> <li>Value of any parameter derived from the outcome measure data (e.g., hazard ratio, mean difference, correlation coefficient)</li> <li>Any of the following, if available: <ul> <li>Confidence Interval</li> <li>Standard deviation or standard error</li> </ul> </li> <li>Additional explanatory comments to interpret the value, if needed: <ul> <li>Directionality of comparison. For subtraction (i.e., A – B or B – A) or a ratio (i.e., A/B or B/A)</li> </ul> </li> </ul> | Estimation Parameter and Value Confidence Interval Parameter Dispersion Estimation Comments |

\*Required

[\*] Conditionally required

Figure 3.30- Statistical Analysis Checklist- Relevant Medication Dosage Decrease

Insert Relevant Medication Dosage Decrease Summary of Results Here



#### Section 4.0: Safety

**Labeling:** The Nu-V3 labeling consists of Instructions for Use and packaging labels. The Instructions for Use include the indications for use; a description of the device, contraindications, warnings, precautions; a list of other devices that are compatible; a detailed summary of the clinical data collected in support of the device; a shelf life; and instructions for the safe use of the device. The labeling satisfies the requirements of 21 CFR 801.109.

Please see the Limitations section above for important warnings and precautions presented in the device labeling.

Risks to Health: Potential unanticipated problems require prompt reporting to Aspire IRB These problems potentially place subjects or others at greater risk of physical or psychological harm than was previously recognized, and warrant consideration of substantive changes in the protocol or informed consent process or other action in order to protect the safety, welfare, or rights of participants. Aspire IRB must be notified within 5 calendar days of the event. The completed IRB Unanticipated Problem form (Appendix 3) must be received by Aspire IRB within 10 calendar days of the event. Unanticipated problems are defined as those problems which alter the risks to subjects or others. This includes any study suspensions or holds. This form will be used to report any problem that is unforeseen or involves risk. One form will be used per event or problem.

| Table 4.1: Unanticipated Problems Involving Risk to Patients or Others | | | |
|---|---|---|---|
| | Phase I | Phase II | Total |
| UPIRTSO 1 (number) | | | |
| UPIRTSO 2 (number) | | | |
| UPIRTSO 3 (number) | | | |
| Overall UPIRTSOs Reported | | | |

| Table 4.2: Risk/ Mitigation Measures | |
|--------------------------------------|---------------------|
| Identified Risk | Mitigation Measures |

Insert Safety Analysis Here



# Section 5.0: Results

**Results:** The principal safety and effectiveness results from patients in the Nu-V3 study are provided below. The primary safety analysis was based on all patients registered and included all reported UPIRTSO events. The primary safety endpoint included imputation for missing clinical outcomes data using the logistic regression method. The imputation model included baseline characteristics including age, sex/gender, marital status, primary language spoken, race/ethnicity, education history, and veteran status.

# **Primary Safety Endpoint:**

Insert Primary Safety Endpoint Statistical Analysis

Insert Primary Safety Endpoint Statistical Table

# **Primary Effectiveness Endpoint:**

Insert Primary Effectiveness Endpoint Statistical Analysis

Insert Primary Effectiveness Endpoint Statistical Table- 8 weeks

### **Secondary Effectiveness Endpoint:**

Insert Primary Effectiveness Endpoint Statistical Analysis

Insert Primary Effectiveness Endpoint Statistical Table: 4, 8, 12 weeks

#### Sub-Analyses:

Insert Sub-Analyses Statistical Analysis

Insert Sub-Analyses Statistical Tables



# **Special Controls:**

Insert Special Control Section Here

# **Benefit/Risk Determination:**

Insert Benefit/Risk Section Here



# **Section 5.0: Administrative Information**

Administrative information consists of the study results point of contact and any agreement between the sponsor and principal investigator (PI) restricting the ability of the PI to discuss the results after the completion of the study.

| Conclusion: | |
|--------------------------|---------------------------------------------------|
| The de novo for Nu-V3 is | and the device is classified under the following: |
| Product Code: | |
| Device Type: | |
| Class: | |
| Regulation: | |